CLINICAL TRIAL: NCT04886934
Title: Open Clinical Investigation to Assess Performance of a Temporary Epicardial Pace Wire With Integrated Sensor for Continuous Postoperative Monitoring of Myocardial Function After Heart Surgery Compared to Ultrasound
Brief Title: Temporary Epicardial Pace Wire With Integrated Sensor for Continuous Postoperative Monitoring of Myocardial Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cardiaccs AS (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-004776-17
Record Dates: First submitted 2021-05-03; First posted 2021-05-14 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Disease; Myocardial Dysfunction
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Safety and clinical performance of the CS1 system (Experimental): Placement of the CS1 device on the left ventricle and externalization of the associated leads through the chest wall during open-heart surgery.
  Interventions: Device: CS1 System

INTERVENTIONS:
Device: CS1 System — Placement of CS1, a temporary bipolar myocardial electrode (TME) with an integrated motion sensor (accelerometer), on the left ventricle and externalization of the associated leads through the chest wall during open-heart surgery. CS1 will remain in place for up to 7 days after surgery and closure of the chest wall.

SUMMARY:
Transesophageal echocardiography is used to monitor cardiac wall motion at various time points during open-heart surgery. After surgery, the measurements are made at various time points by transthoracic echocardiography.

The CS1 system enables continuous, direct measurement of cardiac wall motion. This is achieved through use of temporary pacemaker wires incorporating a motion detector called an accelerometer. Use of TMEs during and after open-heart surgery is part of the normal clinical routine. Continuous monitoring of cardiac wall motion during and after surgery can quickly highlight the need for medical intervention with cardiac drugs and allow very early detection of potentially serious complications leading to abnormal cardiac wall motion.

Cardiac wall motion activity registered by the CS1 system and echocardiography at specific time points during and after surgery will be analyzed to see how well they compare.

DETAILED DESCRIPTION:
Echocardiography is currently the most important and most widely used tool in cardiology besides electrocardiography (ECG). It is reliable for assessing all stages of cardiovascular disease, and it is commonly used to detect heart (cardiac) wall motion dysfunction during and after open-heart surgery.

During open-heart surgery, transesophageal echocardiography (when the echocardiography sensor is introduced into the esophagus) is used to monitor cardiac wall motion at various time points during surgery. After surgery, the measurements are made at various time points by transthoracic echocardiography (when the echocardiography sensor is placed on the chest wall).

Use of the CS1 system enables continuous, direct measurements of cardiac wall motion. This is achieved through use of temporary pacemaker wires (also called temporary myocardial electrodes or TMEs) incorporating a motion detector called an accelerometer. Use of TMEs during and after open-heart surgery is part of the normal clinical routine. Continuous monitoring of cardiac wall motion during the surgery and the post-surgical recovery period can, for example, quickly highlight the need for medical intervention with cardiac drugs and allow very early detection of potentially serious complications such as ischemia (heart muscle is not receiving enough oxygen) and myocardial dysfunction (cardiac wall motion appears abnormal).

The key feature of the CS1 system is that the cardiac wall motion activity registered by the novel TMEs incorporating the accelerometer are displayed visually on a standard medical monitor and synchronized with the patient's ECG data. These data can easily be viewed by medical staff to check if the patient's condition is satisfactory or whether medical intervention is needed.

In the study, the CS1 system will be used in addition to the standard monitoring procedures that include ECG, blood pressures and intermittent echocardiography. Cardiac wall motion activity registered by the CS1 system and echocardiography at specific time points during and after surgery will be analyzed to see how well they compare.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with heart disease requiring surgery
2. Above 18 years
3. Patients suitable for study participation without safety concerns based on the Investigator's evaluation of medical history and physical examination.
4. The patient must be able to understand the aims and objectives of the trial, willing and able to comply with all study related procedures
5. The patient must be willing and able to provide written informed consent prior to participation in the clinical investigation
6. The patient agrees to abstain from enrollment in any other clinical investigation for the duration of the study

Exclusion Criteria:

1. Esophageal disease
2. Atrial fibrillation
3. Pregnancy

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Peak Systolic Velocity (PSV) after increasing heart rate by 25 percent | After surgery: before extubation, while patient is in the intensive care unit (ICU)
  Correlation between relative changes in PSVs measured by CS1 and echocardiography
Change from Baseline PSV after increasing heart rate by 25 percent | After surgery: after extubation and removal of drains, before patient is transferred from ICU to general ward
  Correlation between relative changes in PSVs measured by CS1 and echocardiography

SECONDARY OUTCOMES:
Adverse Events | Up to 30 days after surgery
  Incidence of non-serious and serious adverse events rated for causality
Adverse Device Effects | Up to removal of device at a maximum of 7 days after surgery
  Incidence of non-serious and serious adverse device-related effects
Device Deficiencies | Up to removal of device at a maximum of 7 days after surgery
  Incidence of device deficiencies

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No